CLINICAL TRIAL: NCT03340337
Title: Effects on Isometric Force Induction, Tolerance and Fatigue of Burst-modulated Kilohertz Frequency (Neo-Russian and Aussie) and Low Frequency (Rectangular Biphasic Symmetrical) Neuromuscular Electrical Stimulation in Healthy Subjects
Brief Title: Electrical Stimulation With Different Currents: the Effects on Force, Tolerance and Fatigue in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Universitario de Ciencias de la Salud Fundación H.A. Barceló (Other)
Responsible Party: Principal Investigator, Oscar Ronzio, Professor - Principal Researcher - Member of National Research Committee, Instituto Universitario de Ciencias de la Salud Fundación H.A. Barceló
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RUSSIAN-AUSSIE-RBS-NMES
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: electrical stimulation; Muscle Strength; Fatigue; assessments, pain
MeSH Terms: conditions — Fatigue; Pain

STUDY DESIGN:
Intervention Model Description: Thirty male subjects, right leg dominant, will receive 3 types of electrical stimulation in a randomized order. Aussie current will be delivered by Aussie Sport (Ibramed) device, Neo-Russian by Neurodyn III (Ibramed) device and RBS by a Genesy (Globus) device.
  MVIC and MEIC will be measured with an isometric dynamometer (3 reps x 5 sec work x 120 sec rest). The best rep will be used. Whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum. MVIC will be used for data normalization.
  The VAS will be used to assess tolerance to each treatment. A ratio between MEIC and VAS will be calculated.
  One week later, subjects will receive, ramdomly, a fatigue protocol with the three types of electrical stimulation that consists in 21 reps (5 sec work x 5 sec rest). The data will be normalized with the MVIC and the reps equal or below 50 % of the first rep will be considered as a fatigue rep.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Neo-Russian Electrical Stimulation (Experimental): MVIC will be measured for data normalization. The subjects will receive Neo-Russian electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, the fatigue will be measured with this type of current.
  Interventions: Device: Neo-Russian
- Aussie Electrical Stimulation (Experimental): MVIC will be measured for data normalization. The subjects will receive Aussie electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, the fatigue will be measured with this type of current.
  Interventions: Device: Aussie
- RBS Electrical Stimulation (Experimental): MVIC will be measured for data normalization. The subjects will receive RBS electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, the fatigue will be measured with this type of current.
  Interventions: Device: RBS

INTERVENTIONS:
Device: Neo-Russian — Subjects will receive Neo-Russian electrical stimulation with three reps (5 sec work x 120 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured. They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: Neo-Russian Electrical Stimulation
Device: Aussie — Subjects will receive Aussie electrical stimulation with three reps (5 sec work x 120 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured. They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: Aussie Electrical Stimulation
Device: RBS — Subjects will receive RBS electrical stimulation with three reps (5 sec work x 120 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured. They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: RBS Electrical Stimulation

SUMMARY:
Muscle strength is the amount of force generated by muscle contraction. It could be measured with an isometric dynamometer. This is a validated tool that could be used to measure Maximal Voluntary Isometric Contraction (MVIC) and Maximal Electrical Induced Contraction (MEIC). It is claimed that higher MEIC values will result in more force gained.

If a current is more tolerated it will be easier to achieve better MEIC values. Tolerance to an electrical stimulation could be measured with the Visual Analogue Scale (VAS). A ratio between Normalized MEIC / VAS is often used, implying that the current is better with a higher ratio.

Muscle fatigue is defined as a temporary loss or decrease in force-generating ability due to previous contractions. It is claimed that medium frequency neuromuscular electrical stimulation (NMES) generates more fatigue than low frequency currents.

Aussie is a medium-frequency alternating current, sinusoidal waveform, 1 KHz carrier frequency.

Neo-Russian is a medium-frequency current, rectangular biphasic symmetrical waveform, 2,5 KHz carrier frequency.

Rectangular Biphasic symmetrical (RBS) waveform is a type of Low Pulsed Current (LPC), claimed to be better than classical Russian Current.

Purpose:

As it has been claimed that LPC is better in MEIC and tolerance, the aim of this study is to compare it with two newer medium frequency currents in terms of MEIC, tolerance and fatigue.

Methods:

Thirty male subjects, right leg dominant, will receive randomly the 3 types of electrical stimulation. Before that, the MVIC will be measured for data normalization.

The MVIC and MEIC will be measured with an isometric dynamometer. In both measurements, subjects will be asked to perform three reps (5 sec work x 120 sec rest) and the best one will be used. Whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.

To apply Aussie electrical stimulation, an Aussie Sport (Ibramed) will be used. To apply Neo-Russian, a Neurodyn III (Ibramed) will be used. To apply RBS, a Genesy (Globus) will be used.

The VAS will be used to assess tolerance to each treatment. One week later, the subjects will receive, randomly, a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest) of electrical stimulation with the three types of current. The data will be normalized with the MVIC and the reps equal or below 50 % of the first rep will be considered as a fatigue rep.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Male
* Right leg dominant
* Exercising regularly

Exclusion Criteria:

* History of injuries in the right leg
* Skin lesions
* Having a pacemaker
* Having a cardiovascular disease.
* Having a neurological disorder.
* Exercise 72 h before the procedure.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Born as males.
Enrollment: 30 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar A Ronzio, D.H.Sc, Study Director — Inst. Univer. Fund. H.A. Barceló - U. Maimónides - U. Nac. A. Jauretche
Locations (1):
- Oscar Ronzio, Ciudad Autónoma de Buenos Aire, Buenos Aires F.D., Argentina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sampling: Consecutive non-probability. Population: Students pursuing a degree in Kinesiology and Physiatry at Instituto Universitario de Ciencias de la Salud Fundación H.A. Barceló, at Universidad Maimónides and at Universidad Nacional Arturo Jauretche that met the criteria and accepted to participate.
  Study Start: November 30, 2017 / Study Completion: December 30, 2017
Pre-assignment Details: People that did exercise 72 h before the assignment and procedure were not included.
Groups:
- All Participants: 1. Measurement of MVIC.
  2. All the participants received 3 types of electrical stimulation (Neo-Russian, Aussie and RBS), in a randomized order (balanced permutations, forming 5 x 6 blocks for the three currents).
  3. Determination of Maximal Electrical Induced Contraction (MEIC).
     Dosing information:
     Contraction parameters:
     Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 120 sec Reps: 3, whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.
     Current parameters:
     Neo-Russian: Waveform: Rectangular biphasic symmetrical / Carrier frequency: 2500 Hz / Modulation frequency: 50 Hz / Pulse width: 400 us / Duty cycle: 50 %.
     Aussie: Waveform: Sinousoidal / Carrier frequency: 1000 Hz / Modulation frequency: 50 Hz / Pulse width: 1000 us / Duty cycle: 20 %.
     RBS: Waveform: Rectangular biphasic symmetrical / Frequency: 50 Hz / Pulse width: 400 us.
  4. Washout: 1 week
  5. Fatigue test: All the participants received 3 types of electrical stimulation (Neo-Russian, Aussie and RBS), in a randomized order.
  Dosing information:
  Contraction parameters:
  Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 5 sec Reps: 21. Current parameters: Same as previous.
Period: Overall Study
Arm/Group | All Participants
Started | 30
Received Neo-Russian (All the participants received this type of electrical stimulation, in a randomized order.) | 30
Received Aussie (All the participants received this type of electrical stimulation, in a randomized order.) | 30
Received RBS (All the participants received this type of electrical stimulation, in a randomized order.) | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Maximal Voluntary Isometric Contraction (MVIC) will be measured for data normalization.
  Then, the subjects will receive 3 types of electrical stimulation (Neo-Russian, Aussie and RBS), in a randomized order. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  An isometric dynamometer will be used for acquiring MVIC and MEIC. The protocol will be 3 reps x 5 sec work x 120 sec rest and the best rep will be used. Whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.
  One week later, the subjects will receive a fatigue protocol with the three types of electrical stimulation applied in the randomized order that consists in 21 reps (5 sec work x 5 sec rest). The data will be normalized with the MVIC and the reps equal or below 50 % of the first rep will be considered as a fatigue rep.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (3.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 30
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.71 (1.99)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Voluntary Isometric Contraction (MVIC)
Description: Force generated by the patient during a maximal voluntary isometric contraction, measured by an isometric dynamometer with load cell and computer interface.
  The best of the 3 repetitions was considered. Whenever the third one was the best, additional measurements were taken until a decrease in torque was obtained in order to determine the maximum.
  Unit: Newtons (N)
Time Frame: MVIC was measured at the beggining of the research, on Day 1. Assessed in an average of 7 min
Population: All the participants received 3 types of electrical stimulation (Neo-Russian, Aussie and RBS), in a randomized order, to determine MEIC and Fatigue. As the MVIC was used to normalize "MEIC" and "Fatigue", all study participants were included into one arm.
Measure: Median (Inter-Quartile Range); unit: N
Groups:
- All Study Participants.: As the MVIC was used to normalize the data for others outcome measures, all study participants were included into one arm.
  A short 10-minute walk was taken to warm-up. The patient was positioned in a therapeutic chair with the hip at 110°, stabilizing the trunk (at chest level) and the hip (at the level of the anterior superior iliac spines) with straps. Knee was placed in 90° flexion. A goniometer was used to correctly position the joints at said angles.
  The patient was instructed to cross his arms over his chest and relax. The subject was blindfolded to prevent him from watching the procedure.
  The measuring system was attached to the distal end of the right lower limb by means of an ankle brace.
  The subject was instructed to perform a maximum voluntary isometric contraction.
  Dosing information:
  * Knee angle: 90°
  * Hip angle: 110°
  * Work time: 3 sec
  * Rest time: 120 sec
  * Reps: 3 (Whenever the third one was the best, additional measurements were asked by the software until a decrease in torque was obtained to determine the maximum).
Arm/Group | All Study Participants.
Number analyzed (Participants) | 30
N | 419.68 [299.51 to 531.77]

2. Primary Outcome: Maximal Electrical Induced Contraction (MEIC)
Description: Force generated in the muscle while applying electrical stimulation, measured by an isometric dynamometer with load cell and computer interface. This data (in Newtons) was normalized with the MVIC.
  Unit: percentage of MVIC
Time Frame: MEIC was measured on Day 1. Order: MVIC - Rest: 120 sec. - MEIC current 1 - Rest: 120 sec. - MEIC current 2 - Rest: 120 sec. - MEIC current 3 - Rest: 120 sec. - Assessed in an average of 21 min.
Measure: Median (Inter-Quartile Range); unit: percentage of MVIC
Groups:
- Neo-Russian Electrical Stimulation: After measuring the MVIC, subject rested for 120 seconds (while searching for motor points for rectus femoris and vastus medialis).
  All subjects received all currents in a randomized order. The subject was asked not to make any voluntary contraction. Neo-Russian electrical stimulation was applied. At the higher tolerated intensity, the MEIC was measured and normalized with the MVIC.
  Dosing information:
  * Knee angle: 90°
  * Hip angle: 110°
  Contraction parameters:
  Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 120 sec Reps: 3, whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.
  Current parameters:
  Neo-Russian: Waveform: Rectangular biphasic symmetrical / Carrier frequency: 2500 Hz / Modulation frequency: 50 Hz / Pulse width: 400 us / Duty cycle: 50 %.
  An interval of 120 seconds was also taken between the determinations of the MEIC with each current, in order to minimize fatigue.
- Aussie Electrical Stimulation: After measuring the MVIC, subject rested for 120 seconds (while searching for motor points for rectus femoris and vastus medialis).
  All subjects received all currents in a randomized order. The subject was asked not to make any voluntary contraction. Aussie electrical stimulation was applied. At the higher tolerated intensity, the MEIC was measured and normalized with the MVIC.
  Dosing information:
  * Knee angle: 90°
  * Hip angle: 110°
  Contraction parameters:
  Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 120 sec Reps: 3, whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.
  Current parameters:
  Aussie: Waveform: Sinousoidal / Carrier frequency: 1000 Hz / Modulation frequency: 50 Hz / Pulse width: 1000 us / Duty cycle: 20 %.
  An interval of 120 seconds was also taken between the determinations of the MEIC with each current, in order to minimize fatigue.
- RBS Electrical Stimulation: After measuring the MVIC, subject rested for 120 seconds (while searching for motor points for rectus femoris and vastus medialis).
  All subjects received all currents in a randomized order. The subject was asked not to make any voluntary contraction. RBS electrical stimulation was applied. At the higher tolerated intensity, the MEIC was measured and normalized with the MVIC.
  Dosing information:
  * Knee angle: 90°
  * Hip angle: 110°
  Contraction parameters:
  Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 120 sec Reps: 3, whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.
  Current parameters:
  RBS: Waveform: Rectangular biphasic symmetrical / Frequency: 50 Hz / Pulse width: 400 us.
  An interval of 120 seconds was also taken between the determinations of the MEIC with each current, in order to minimize fatigue.
Arm/Group | Neo-Russian Electrical Stimulation | Aussie Electrical Stimulation | RBS Electrical Stimulation
Number analyzed (Participants) | 30 | 30 | 30
percentage of MVIC | 30.30 [12.23 to 53.22] | 13.44 [8.66 to 37.00] | 10.05 [4.86 to 25.25]

3. Primary Outcome: Visual Analogue Scale (VAS)
Description: Visual Analogue Scale (VAS): Magnitude of pain, marked in a analogue scale by participants, to determine how unpleasant was each type of electrical stimulation (applied in randomized order). Expresed in centimeters.
  * Minimum value: 0
  * Maximum value: 10
  * A higher score implicates a worse outcome. VAS was evaluated 3 times, 1 per type of electrical stimulation.
Time Frame: Asked after evaluation of MEIC wiht each type of current. VAS current 1 - VAS current 2 - VAS current 3 - Assessed in average of 15 seconds for each current.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neo-Russian Electrical Stimulation: After recording the MEIC of Neo-Russian electrical stimulation, the subject was given a VAS and was asked to indicate how unpleasant he found the electro-stimulation with this current, with 0 (on the left) being "no pain" and 10 (on the right) the equivalent of "crying in pain".
- Aussie Electrical Stimulation: After recording the MEIC of Aussie electrical stimulation, the subject was given a VAS and was asked to indicate how unpleasant he found the electro-stimulation with this current, with 0 (on the left) being "no pain" and 10 (on the right) the equivalent of "crying in pain".
- RBS Electrical Stimulation: After recording the MEIC of RBS electrical stimulation, the subject was given a VAS and was asked to indicate how unpleasant he found the electro-stimulation with this current, with 0 (on the left) being "no pain" and 10 (on the right) the equivalent of "crying in pain".
Arm/Group | Neo-Russian Electrical Stimulation | Aussie Electrical Stimulation | RBS Electrical Stimulation
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 5.54 (2.26) | 6.20 (2.57) | 5.15 (2.59)

4. Secondary Outcome: Fatigue
Description: Number of repetitions, while applying electrical stimulation, equal to or lower than 50% of the first of 21 reps, previously normalized with MVIC Units: units on scale. Range: from 0 to 21. A higher value represents a worse outcome.
Time Frame: Washout: 1 Week. Fatigue current 1 - Rest: 120 sec. - Fatigue current 2 - Rest: 120 sec. - Fatigue current 3 - Assessed in an average of 21 min.
Measure: Median (Inter-Quartile Range); unit: repetitions
Groups:
- Neo-Russian Electrical Stimulation: Fatigue induced by the electrical stimulation was measured in a randomized order after one week of washout period.
  An isometric dynamometer was used. The patient was instructed to cross his arms over his chest, to relax and not to make any voluntary contraction. The subject was blindfolded to prevent him from watching the procedure. The measuring system was attached to the distal end of the right lower limb.
  The intensity was increased until it reached the maximum tolerable by the subject. Data was taken from the MEIC of 21 contractions.
  Each repetition was normalized as a percentage of MVIC. Then, Repetition 1 was considered to be 100 %. Subsequently, it was calculated what percentage of repetition 1 the subsequent repetitions corresponded to. The number of repetitions equal to or lower than 50% was then counted, thus determining the fatigue induced by each type of electrical stimulation.
  An interval of 120 seconds was also taken between the determinations of the Fatigue test with each current.
  Dosing information:
  * Knee angle: 90°
  * Hip angle: 110°
  Contraction parameters:
  Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 5 sec Reps: 21 Neo-Russian: Waveform: Rectangular biphasic symmetrical / Carrier frequency: 2500 Hz / Modulation frequency: 50 Hz / Pulse width: 400 us / Duty cycle: 50 %.
- Aussie Electrical Stimulation: Fatigue induced by the electrical stimulation was measured in a randomized order after one week of washout period.
  An isometric dynamometer was used. The patient was instructed to cross his arms over his chest, to relax and not to make any voluntary contraction. The subject was blindfolded to prevent him from watching the procedure. The measuring system was attached to the distal end of the right lower limb.
  The intensity was increased until it reached the maximum tolerable by the subject. Data was taken from the MEIC of 21 contractions.
  Each repetition was normalized as a percentage of MVIC. Then, Repetition 1 was considered to be 100 %. Subsequently, it was calculated what percentage of repetition 1 the subsequent repetitions corresponded to. The number of repetitions equal to or lower than 50% was then counted, thus determining the fatigue induced by each type of electrical stimulation.
  An interval of 120 seconds was also taken between the determinations of the Fatigue test with each current.
  Dosing information:
  * Knee angle: 90°
  * Hip angle: 110°
  Contraction parameters:
  Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 5 sec Reps: 21 Aussie: Waveform: Sinousoidal / Carrier frequency: 1000 Hz / Modulation frequency: 50 Hz / Pulse width: 1000 us / Duty cycle: 20 %.
- RBS Electrical Stimulation: Fatigue induced by the electrical stimulation was measured in a randomized order after one week of washout period.
  An isometric dynamometer was used. The patient was instructed to cross his arms over his chest, to relax and not to make any voluntary contraction. The subject was blindfolded to prevent him from watching the procedure. The measuring system was attached to the distal end of the right lower limb.
  The intensity was increased until it reached the maximum tolerable by the subject. Data was taken from the MEIC of 21 contractions.
  Each repetition was normalized as a percentage of MVIC. Then, Repetition 1 was considered to be 100 %. Subsequently, it was calculated what percentage of repetition 1 the subsequent repetitions corresponded to. The number of repetitions equal to or lower than 50% was then counted, thus determining the fatigue induced by each type of electrical stimulation.
  An interval of 120 seconds was also taken between the determinations of the Fatigue test with each current.
  Dosing information:
  * Knee angle: 90°
  * Hip angle: 110°
  Contraction parameters:
  Ramp-up: 1 sec On time: 3 sec Ramp-down: 1 sec Total work time: 5 sec Rest time: 5 sec Reps: 21 RBS: Waveform: Rectangular biphasic symmetrical / Frequency: 50 Hz / Pulse width: 400 us.
Arm/Group | Neo-Russian Electrical Stimulation | Aussie Electrical Stimulation | RBS Electrical Stimulation
Number analyzed (Participants) | 30 | 30 | 30
repetitions | 6.5 [0.00 to 11.50] | 3.00 [0.00 to 12.25] | 0.00 [0.00 to 0.00]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Participant were asked if they experiment delayed onset muscle soreness (DOMS) or any other kind of pain.
Groups:
- Neo-Russian Electrical Stimulation: MVIC was measured for data normalization.
  Subjects received Neo-Russian electrical stimulation with three reps (5 sec work x 120 sec rest), and the Maximal Electrical Induced Contraction (MEIC) was measured.
  They were asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects received a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) was measured for each contraction.
- Aussie Electrical Stimulation: MVIC was measured for data normalization.
  Subjects received Aussie electrical stimulation with three reps (5 sec work x 120 sec rest), and the Maximal Electrical Induced Contraction (MEIC) was measured.
  They were asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects received a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) was measured for each contraction.
- RBS Electrical Stimulation: MVIC was measured for data normalization.
  Subjects received RBS electrical stimulation with three reps (5 sec work x 120 sec rest), and the Maximal Electrical Induced Contraction (MEIC) was measured.
  They were asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects received a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) was measured for each contraction.
Arm/Group | Neo-Russian Electrical Stimulation | Aussie Electrical Stimulation | RBS Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03340337/Prot_SAP_000.pdf